CLINICAL TRIAL: NCT06050967
Title: A Feasibility Open-labeled Clinical Trial Using a Second-generation Artificial Intelligence-based Therapeutic Regimen in Patients With Gaucher Disease Treated With Enzyme Replacement Therapy
Brief Title: A Second-generation AI Based Therapeutic Regimen in Patients With Gaucher Disease Treated With Enzyme Replacement Therapy.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0056-21-SZMC
Record Dates: First submitted 2023-09-01; First posted 2023-09-22 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-08

CONDITIONS: Gaucher Disease Type 1
MeSH Terms: conditions — Gaucher Disease | interventions — Enzyme Replacement Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- individualized treatment plan with random dosage and time of administration (Experimental): Baseline clinical and laboratory parameters acquired at the screening included: a physical examination, complete blood count (CBC), Lyso-GB1 , and a 36-item short-form survey (SF-36) for quality-of-life examination. Once providing informed consent, the Altus Care™ application was installed on the patient's cellular phone. In coordination with the patient's treating physician and the home treating nurse5 , an individualized treatment plan was prepared for each patient within a pre-defined range of minimal and maximal once in two weeks ERT dosages and timing frames for its administration. Per protocol, the patient's monthly dose wasn't changed, but each dose and the timing of administration was changed randomly using the app.
  Interventions: Combination Product: Enzyme replacement therapy for Gaucher disease in combination with altus care application

INTERVENTIONS:
Combination Product: Enzyme replacement therapy for Gaucher disease in combination with altus care application — In coordination with the patient's treating physician and the home treating nurse, an individualized treatment plan was prepared for each patient within a pre-defined range of minimal and maximal once in two weeks enzyme replacement therapy dosages and timing frames for its administration. Per protocol, the patient's monthly dose was not changed, but each dose and the timing of administration was changed randomly using the app.

SUMMARY:
An open-labeled, prospective, single-center proof-of-concept study. Patients with Gaucher Disease aged 18-75 who received intravenous Enzyme Replacement Therapy once every two weeks were enrolled. The study utilized the Altus Care™ cellular phone-based application, which integrated an algorithm-based approach to provide random dosing regimens within a pre-defined range determined by the physician. The app allowed personalized therapeutic regimens with variations in dosages and administration times.

DETAILED DESCRIPTION:
Patients diagnosed with GD and intravenously treated at home with a regular dose of Enzyme Replacement Therapy once every two weeks for 6 months (30- 60 U/kg per mouth) were included in the study.

We installed Altus Care™- this is a cellular phone-based application that allows easy digitization of treatment plans or research protocols and remote implementation. In coordination with the patient's treating physician and the home treating nurse, an individualized treatment plan was prepared for each patient within a pre-defined range of minimal and maximal once in two weeks ERT dosages and timing frames for its administration. Per protocol, the patient's monthly dose was not changed, but each dose and the timing of administration was changed randomly using the app.

During the follow-up period, the research coordinator made a regular weekly checkup by phone, questioning the patient's clinical well-being and adherence to the treatment plan. A physical examination, CBC, and Lyso-GB1 assessed response to therapy were done approximately every two months (twice during the study and once again at the end of the follow-up). The patients filled out SF-36 questionnaires at the beginning and the end of the follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Adult >18 years old
* Non-pregnant
* Diagnosed with Gaucher disease
* Treated with ERT for a minimum of 3 years
* An unchanged dose in the past 6/12 months

Exclusion Criteria:

* Pregnant
* Patients with evidence of severe infectious, malignant, autoimmune, or other disabling systemic diseases
* Patients unable to provide written informed consent
* Patients that do not possess a smartphone
* Patients who cant adhere to the visit schedule and protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Platelet | 6 month
  number of platelets per L. normal range 150,000 to 450,000. In Gaucher disease lower platelets means higher disease activity
Hemoglobin | 6 month
  Hemoglobin concentration in gram/dl. normal range 13.8 to 17.2 for males and 12.1 to 15.1 for females. The lower the hemoglobin the higher Gaucher disease activity
Lyso GB1 | 6 month
  Lyso GB1 level in ng/ml. For healthy individuals the levels should be trace less than 4.9ng/ml. In patients with Gaucher disease the higher the level the higher the disease activity.
SF-36 | 6 month
  score of 0-100. 0 means worse and 100 means best.

CONTACTS AND LOCATIONS:
Overall Officials: Noa Hurvitz, MD, Principal Investigator — Faculty of Medicine, Hebrew University, Jerusalem, Israel.
Locations (1):
- Hebrew university, Jerusalem, Israel